CLINICAL TRIAL: NCT06857890
Title: An Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of the Drug Grammidin With Anesthetic, a Metered Dose Topical Spray Following Single Administration in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetic Profile of Grammidin With Anesthetic, a Metered Dose Topical Spray in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRM-01-07-2024
Record Dates: First submitted 2025-02-17; First posted 2025-03-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Gramicidin; Cetylpyridinium; benoxinate; Anesthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT sequence: Grammidin with anesthetic neo followed by Grammidin with anesthetic (Experimental): RT sequence where R is Grammidin with anesthetic neo, lozenges, and T is Grammidin with anesthetic, a metered dose topical spray
  Interventions: Drug: Grammidin with anesthetic neo; Drug: Grammidin with anesthetic, a metered dose topical spray
- TR sequence: Grammidin with anesthetic followed by Grammidin with anesthetic neo (Experimental): TR sequence where T is Grammidin with anesthetic, a metered dose topical spray, and R is Grammidin with anesthetic neo, lozenges
  Interventions: Drug: Grammidin with anesthetic neo; Drug: Grammidin with anesthetic, a metered dose topical spray

INTERVENTIONS:
Drug: Grammidin with anesthetic neo — Grammidin with anesthetic neo, lozenges, 1 lozenge to be taken once under fed conditions.
  Other Names: gramicidin s; cetylpyridinium chloride; oxybuprocaine
Drug: Grammidin with anesthetic, a metered dose topical spray — Grammidin with anesthetic, a metered dose topical spray, 4 sprays to be taken once under fed conditions
  Other Names: gramicidin s; cetylpyridinium chloride; oxybuprocaine

SUMMARY:
This study aims to evaluate the safety, tolerability, and pharmacokinetic profile of the Grammidin with anesthetic, a metered dose topical spray, compared to Grammidin with anesthetic neo, lozenges following single administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily and personally signed informed consent form by a healthy volunteer obtained prior to the conduct of any study-related procedure;
2. Males and females aged 18 to 45 years (inclusive);
3. Verified healthy status as demonstrated by the absence of clinically significant abnormalities in medical history, physical examination, laboratory tests, and other diagnostic procedures specified in the protocol;
4. Blood pressure (BP) level: systolic blood pressure (SBP) from 99 to 129 mm Hg (inclusive), diastolic blood pressure (DBP) from 70 to 89 mm Hg (inclusive);
5. Heart rate (HR) from 60 to 89 beats per minute (inclusive);
6. Respiratory rate (RR) from 12 to 20 breaths per minute (inclusive);
7. Body temperature from 36.0°C to 36.9°C (inclusive);
8. Body mass index (BMI) between 18.5 kg/m² and 30 kg/m², with a minimum body weight of ≥ 55 kg for men and ≥ 45 kg for women;
9. Consent to use adequate contraceptive methods throughout the study and for 30 days after its completion, with a negative urine pregnancy test result for women of childbearing potential.

Non-Inclusion Criteria:

1. Clinically significant allergic history;
2. Hypersensitivity to active and/or excipient substances in the investigational drug and comparator drug in the medical history;
3. Drug intolerance to active and/or excipient substances in the investigational drug and comparator drug in the medical history;
4. Chronic diseases of the kidneys, liver, gastrointestinal tract (GIT), cardiovascular, lymphatic, respiratory, nervous, endocrine, musculoskeletal, urogenital, and immune systems, as well as skin, hematopoietic organs, and the eye;
5. Erosive-ulcerative lesions of the oral mucosa (aphthous stomatitis, mechanical trauma due to dental diseases, herpes lesions, and any other condition resulting in compromised integrity of the oral mucosa);
6. Surgical interventions on the GIT in the medical history (except for appendectomy performed at least 1 year prior to screening);
7. Diseases/conditions that, in the investigator's judgment, may affect the absorption, distribution, metabolism, or excretion of the investigational drugs;
8. Acute infectious diseases less than 4 weeks before screening;
9. Use of medications (drugs) that significantly affect hemodynamics and drugs affecting liver function (barbiturates, omeprazole, cimetidine, etc.) less than 2 months before screening;
10. Regular use of medications less than 2 weeks before screening and single use of medications less than 7 days before screening (including over-the-counter medications, vitamins, dietary supplements, herbal medicines);
11. Blood or plasma donating within 3 months prior to screening;
12. Use of hormonal contraceptives (in women) within 2 months prior to screening;
13. Use of depot injections of any medications within 3 months prior to screening;
14. Pregnancy or lactation; positive urine pregnancy test result for women of childbearing potential;
15. Female subjects of childbearing potential who had unprotected sexual intercourse with an unsterilized male partner within 30 days prior to administration investigational drugs;
16. Participation in another clinical study within 3 months prior to screening or concurrently with this study;
17. Consumption of more than 10 alcohol units per week (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of wine, or 50 ml of strong alcoholic beverages) in the last month before inclusion in the study or a history of alcoholism, drug addiction, or substance abuse;
18. Smoking more than 10 cigarettes per day currently or smoking that amount in the past 6 months prior to screening; unwillingness to refrain from smoking during hospitalization;
19. Consumption of alcohol, caffeine, and xanthine-containing products within 7 days prior to taking investigational drugs;
20. Consumption of citrus fruits, cranberries, rose hips and products containing them, or preparations/products containing St. John's wort within 7 days prior to taking investigational drugs;
21. Dehydration due to diarrhea, vomiting, or other causes within the last 24 hours prior to taking investigational drugs;
22. Positive blood test for antibodies to human immunodeficiency virus (HIV) types 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens during screening;
23. Positive rapid test for SARS-CoV-2 at screening;
24. ECG abnormalities in medical history and/or during screening;
25. Positive urine test for narcotic substances and potent medications during screening;
26. Positive breath alcohol test result during screening;
27. Planning hospitalization during the study period for any reason other than hospitalization specified in this protocol;
28. Inability or unwillingness to comply with protocol requirements, perform procedures prescribed by the protocol, or adhere to dietary and activity restrictions;
29. Membership in a vulnerable population? including but not limited to students of medical, pharmaceutical and dental educational institutions, junior staff of clinics and laboratories, employees of pharmaceutical companies, military personnel, prisoners, residents of care facillities, individuals with low income or unemployed, members of ethnic minorities, homeless persons, vagrants, refugees, individuals under guardianship or conservatorship, ndividuals unable to provide informed consent and law enforcement personnel;
30. Dental procedures performed within 3 weeks prior to screening;
31. Other conditions that in the judgment of the Investigator may prevent volunteer inclusion in the study or lead to premature withdrawal from the study including adherence to fasting or special diets (e.g., vegetarianism, veganism, salt restriction) or special lifestyles (night work, extreme physical exertion).

Exclusion Criteria:

1. Withdrawal of the volunteer from further participation in the study;
2. Non-compliance by the volunteer with the study participation rules (missed study procedures, self-administration of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Emergence of reasons/situations during the study that threaten the safety of the volunteer (e.g., hypersensitivity reactions, etc.);
4. Volunteers selected for participation in the study who do not meet inclusion/exclusion criteria;
5. Development of a severe adverse event (SAE) in the volunteer during the study;
6. The volunteer undergoes or requires treatment that may affect the pharmacokinetic parameters (PKP) of the investigational drugs;
7. Missed collection of 2 or more consecutive blood samples or 3 or more blood samples within one study period;
8. Occurrence of vomiting/diarrhea within 6 hours after taking the investigational drug;
9. Positive urine test for narcotic substances and potent medications;
10. Positive breath test for alcohol vapors;
11. Positive pregnancy test result in women;
12. Positive SARS-CoV-2 test result;
13. Emergence of other reasons during the study that prevent conducting the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 24 hours after each drug intake.
  Maximum plasma concentration (Cmax) of gramicidin S, oxybuprocaine hydrochloride, and cetylpyridinium chloride. The same analytes would be used for other pharmacokinetic measures listed below.
Pharmacokinetics - tmax | From 0 to 24 hours after each drug intake.
  Time to reach Cmax (tmax)
Pharmacokinetics - AUC0-t | From 0 to 24 hours after each drug intake.
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t)
Pharmacokinetics - AUC0-inf | From 0 hours after each drug intake (extrapolated to infinity)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf)
Pharmacokinetics - AUCextr | From 0 hours after each drug intake (extrapolated to infinity)
  Extrapolated AUC defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - t1/2 | From 0 to 24 hours after each drug intake.
  Elimination half-life (t1/2)
Pharmacokinetics - kel | From 0 to 24 hours after each drug intake.
  Elimination constant (kel)
Pharmacokinetics - MRT | From 0 to 24 hours after each drug intake.
  Mean residence time (MRT)
Pharmacokinetics - Vd | From 0 to 24 hours after each drug intake.
  Volume of distribution
Pharmacokinetics - CL | From 0 to 24 hours after each drug intake.
  Clearance (CL)
Pharmacokinetics - number of terminal timepoints | From 0 to 24 hours after each drug intake.
  Number of points in the terminal logarithmic phase used to estimate the terminal elimination rate constant

SECONDARY OUTCOMES:
Adverse event type | From screeninig (days -14 to -1) to the end of study (day 15 ± 1)
  Adverse events will be assessed by complaints, results of physical examination, results of heart rate and blood pressure assessment, results of respiratory rate assessment, body temperature, laboratory monitoring (clinical blood count, biochemical blood count, urinalysis), electrocardiography; adverse events will be classified in accordance to MedDRA.
Adverse event number | From screeninig (days -14 to -1) to the end of study (day 15 ± 1)
  Number of adverse events registered during the study
Adverse event severety | From screeninig (days -14 to -1) to the end of study (day 15 ± 1)
  Severity of adverse events registered during the study
Drop-outs associated with adverse events | From screeninig (days -14 to -1) to the end of study (day 15 ± 1)
  The number of cases of early termination of participation in the study due to the development of adverse events and/or serious adverse events associated with the study drug
Safety and Tolerability: volunteer complaints | From screeninig (days -14 to -1) to the end of study (day 15 ± 1)
  Description of complaints, recieved from volunteer
Safety and Tolerability: physical examination results - cardiovascular system | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the cardiovascular system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - respiratory system | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the respiratory system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - digestive tract | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the digestive tract on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - endocrine system | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the endocrine system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - musculoskeletal system | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the musculoskeletal system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - nervous system | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the nervous system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - sensory systems | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the sensory systems on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - skin/visible mucous membranes | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  An assessment of the condition of the skin/visible mucous membranes on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: vital signs - systolic blood pressure | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  Systolic blood pressure (SBP, mmHg)
Safety and Tolerability: vital signs - diastolic blood pressure | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  Diastolic blood pressure (DBP, mmHg)
Safety and Tolerability: vital signs - heart rate | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  Heart rate (HR, bpm)
Safety and Tolerability: vital signs - body temperature (Celsius temperature scale) | Screeninig (days -14 to -1), day -1 to 2, day 7 to 9, day 15 ± 1
  Body temperature (Celsius temperature scale)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screeninig (days -14 to -1), day 1, 2, 8, 9, 15 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screeninig (days -14 to -1), day 1, 2, 8, 9, 15 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: PQ interval (is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screeninig (days -14 to -1), day 1, 2, 8, 9, 15 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: QRS complex (the QRS complex is the combination of three of the graphical deflections seen on a typical electrocardiogram)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval | Screeninig (days -14 to -1), day 1, 2, 8, 9, 15 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: corrected QT interval (distance from the beginning of the QRS complex to the end of the T wave)
Safety and Tolerability: clinical blood test - hemoglobin | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Hemoglobin (g/L)
Safety and Tolerability: clinical blood test - hematocrit | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Hematocrit (%)
Safety and Tolerability: clinical blood test - red blood cell count | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Red blood cell count (cells/L)
Safety and Tolerability: clinical blood test - platelet count | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Platelet count (cells/L)
Safety and Tolerability: clinical blood test - leukocyte count | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte count (cells/L)
Safety and Tolerability: clinical blood test - erythrocyte sedimentation rate | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Erythrocyte sedimentation rate (mm/h)
Safety and Tolerability: clinical blood test - myelocytes | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (myelocytes, %)
Safety and Tolerability: clinical blood test - band neutrophils | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (band neutrophils, %)
Safety and Tolerability: clinical blood test - segmented neutrophils | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (segmented neutrophils, %)
Safety and Tolerability: clinical blood test - eosinophils | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (eosinophils, %)
Safety and Tolerability: clinical blood test - basophils | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (basophils, %)
Safety and Tolerability: clinical blood test - monocytes | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (monocytes, %)
Safety and Tolerability: clinical blood test - lymphocytes | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Leukocyte formula (lymphocytes, %)
Safety and Tolerability: urinalysis - specific gravity | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Protein concentration (g/L)
Safety and Tolerability: urinalysis - glucose | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Glucose concentration (mmol/L)
Safety and Tolerability: urinalysis - red blood cells | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Red blood cell content (number in sight)
Safety and Tolerability: urinalysis - white blood cells | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  White blood cell content (number in sight)
Safety and Tolerability: urinalysis - epithelial cells | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Epithelial cell content (number in sight)
Safety and Tolerability: urinalysis - casts | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Presence of casts (Yes/No)
Safety and Tolerability: urinalysis - mucus | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Presence of mucus (Yes/No)
Safety and Tolerability: urinalysis - bacteria | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Presence of bacteria (Yes/No)
Safety and Tolerability: urinalysis (microscopy) | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Microscopy of urine sediment is performed if it is present
Safety and Tolerability: blood chemistry - glucose | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Glucose concentration (mmol/L)
Safety and Tolerability: blood chemistry - cholesterol | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Total cholesterol concentration (mmol/L)
Safety and Tolerability: blood chemistry - protein | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Total protein concentration (g/L)
Safety and Tolerability: blood chemistry - bilirubin | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Total bilirubin concentration (micromol/L)
Safety and Tolerability: blood chemistry - creatinine | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Creatinine concentration (micromol/L)
Safety and Tolerability: blood chemistry - alkaline phosphatase | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Alkaline phosphatase activity (U/L)
Safety and Tolerability: blood chemistry - alanine transaminase | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Alanine transaminase activity (U/L)
Safety and Tolerability: blood chemistry - aspartate transaminase | Screeninig (days -14 to -1), day 2, 9, 15 ± 1
  Aspartate transaminase activity (U/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Separate Medical Unit "CoMed" (LLC "Ligand Research"), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No